CLINICAL TRIAL: NCT06501404
Title: Effects of Probiotic Supplementation During the Neonatal Period on the Preterm Infant
Brief Title: PREMAPROB. Probiotics to Prevent Necrotizing Enterocolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José Antonio Hurtado Suazo (Other)
Collaborators: University Hospital Virgen de las Nieves (Other); Hospital Regional de Malaga (Other); Hospital of Jaen (Other); Hospital Costa del Sol (Other); Hospital Universitario Torrecárdenas (Other); Hospital Universitario Virgen Macarena (Other); Complejo Hospitalario de Especialidades Juan Ramón Jimenez (Other); Hospital Universitario de Valme (Other); Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Puerta del Mar (Other); Hospital General Universitario Santa Lucia (Other); Hospital del SAS de Jerez (Other)
Responsible Party: Sponsor-Investigator, José Antonio Hurtado Suazo, Head of Neonatolgy Division. University Hospital Virgen de las Nieves, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Organization: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PN01
Record Dates: First submitted 2024-06-19; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Premature Infants; Necrotizing Enterocolitis
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose of probiotic mixture (Experimental): A daily high dose of a mixture of probiotics (Lactobacillus Fermentum CECT 5716 and Bifidobacterium breve CECT 7263), was given orally starting in the first 72 hours of life, until 36+6 weeks of postmenstrual age or discharge The total dose was 1x109 CFU of each of the strains
  Interventions: Dietary Supplement: High dose group
- Low dose of probiotic mixture (Experimental): A daily low dose of a mixture of probiotics (Lactobacillus Fermentum CECT 5716 and Bifidobacterium breve CECT 7263), was given orally starting in the first 72 hours of life, until 36+6 weeks of postmenstrual age or discharge The total dose was 1x106 CFU of each of the strains
  Interventions: Dietary Supplement: Low dose group

INTERVENTIONS:
Dietary Supplement: High dose group — A daily high dose of a mixture of probiotics (Lactobacillus Fermentum CECT 5716 and Bifidobacterium breve CECT 7263), was given orally starting in the first 72 hours of life, until 36+6 weeks of postmenstrual age or discharge The total dose was 1x109 CFU of each of the strains
  Arms: High dose of probiotic mixture
Dietary Supplement: Low dose group — A daily low dose of a mixture of probiotics (Lactobacillus Fermentum CECT 5716 and Bifidobacterium breve CECT 7263), was given orally starting in the first 72 hours of life, until 36+6 weeks of postmenstrual age or discharge The total dose was 1x106 CFU of each of the strains
  Arms: Low dose of probiotic mixture

SUMMARY:
The main objective of this study is to assess the impact of two different doses of a mixture of probiotics from two strains isolated in human milk on the incidence of severe necrotizing enterocolitis (NEC) and death among preterm infants of gestational age less than or equal to 32 weeks of gestation and weighing between 750 and 1500 g.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants of gestational age less than 33 weeks of gestation with birth weight below 1500 g, admitted to the Neonatology Unit.
* Premature newborns who meet the above criteria and receive enteral feeding (mother breast milk, donors milk and/or premature formula) from the amount of 5 ml/kg/day.

Exclusion Criteria:

* Any clinical circumstance that prevents the initiation of enteral nutrition in the first 72 hours of life.
* Chromosomopathies and complex fetal malformations, incompatible with enteral nutrition in the first 72 hours of life.
* Non-acceptance of informed consent to participate in the study by the parents or legal guardians of the newborn.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 583 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of necrotizing enterocolitis and all-cause mortality | From birth until three months
  The primary objective of the study was to determine the incidence of necrotizing enterocolitis (modified Bell classification stages II and III) and all-cause mortality during hospital stay in both intervention groups.

SECONDARY OUTCOMES:
Intestinal colonization by administered strains | From birth until three months
Incidence of Late Onset Sepsis | From birth until three months
  Incidence of Late Onset Sepsis. In accordance with the criteria used by the Castrillo Group for neonatal infections in Spain (compatible clinical symptoms, elevation of water-phase reactants and positive blood culture)
Time to complete enteral nutrition | From birth until three months
  Time to reach complete enteral nutrition 140 ml/kg/day
Days of Central Vascular Catheter | From birth until three months
Length of hospital stay | From birth until three months
  Days of hospital stay
Weight change | From birth until three months
Incidence of Bronchopulmonary Dysplasia | From birth until three months
Incidence of patent ductus arteriosus | From birth until three months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Virgen de las Nieves, Granada, Spain

IPD SHARING:
Plan to Share IPD: No